CLINICAL TRIAL: NCT04817254
Title: Phase II Trial Evaluating the Association of Peripheral Blood Immunologic Response to Therapeutic Response to Adjuvant Treatment With Immune Checkpoint Inhibition (ICI) in Patients With Newly Diagnosed Glioblastoma or Gliosarcoma
Brief Title: Association of Peripheral Blood Immunologic Response to Therapeutic Response to Adjuvant Treatment With Immune Checkpoint Inhibition (ICI) in Patients With Newly Diagnosed Glioblastoma or Gliosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210015; 21-C-0015
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12-19

CONDITIONS: Glioblastoma; Gliosarcoma; Malignant Glioma
Keywords: Brain Cancer; Quality of Life
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Nivolumab + Ipilimumab 1mg/kg + TMZ
  Interventions: Drug: TMZ; Drug: Nivolumab; Drug: ipilimumab 1mg/kg
- Arm 2 (Experimental): Nivolumab + Ipilimumab 3mg/kg + TMZ
  Interventions: Drug: TMZ; Drug: ipilimumab 3mg/kg; Drug: Nivolumab

INTERVENTIONS:
Drug: TMZ — 150 mg/m2 on days 1-5 of cycles 1-6
Drug: ipilimumab 3mg/kg — 3 mg/kg q 4 weeks for cycles 1-4
  Arms: Arm 2
Drug: Nivolumab — 1 mg/kg IV q2weeks for cycles 1-4, then 480 mg q 4 weeks for cycles 5-16
Drug: ipilimumab 1mg/kg — 1 mg/kg q 4 weeks for cycles 1-4
  Arms: Arm 1

SUMMARY:
Background:

Glioblastoma (GBM) is a type of malignant glioma. These cancers are nearly always fatal. People who develop these cancers get aggressive treatments. But the tumors almost always recur. Researchers want to study people with newly diagnosed disease to learn more.

Objective:

To study people with newly diagnosed GBM or gliosarcoma to look at the changes in immune cells in the blood of those who take ipilimumab and nivolumab, along with temozolomide.

Eligibility:

Adults ages 18 and older with newly diagnosed GBM or gliosarcoma, who have had surgical removal of their tumor and have completed standard initial chemotherapy and radiation therapy.

Design:

Participants will be screened with the following:

Medical record review

Medical history

Physical exam

Tests to assess their nervous system and their ability to do typical activities

Blood tests

Tumor assessment. For this, they will have magnetic resonance imaging (MRI). They may get a contrast dye through an intravenous (IV) catheter. The MRI scanner makes noise. They will get earplugs.

Electrocardiogram. It measures heart rate and rhythm. They will lie still. Sticky pads will be placed on their chest, arms, and legs.

Screening tests will be repeated during the study.

Treatment will be given in cycles. Each cycle lasts 4 weeks. Participants will get nivolumab and ipilimumab via IV. They will take temozolomide by mouth. They will keep a pill diary.

Participants will fill out surveys about their symptoms.

Participants will have follow-up visits about 60 days and 100 days after treatment ends. Then they will be contacted every 6 months for the rest of their life.

DETAILED DESCRIPTION:
Background:

Glioblastoma (GBM) represents an aggressive malignancy with limited therapeutic options. The immunosuppressive nature of GBM may be reversible with immune checkpoint inhibitor (ICI) treatment, however, initial studies have yet to demonstrate this. It is postulated that trafficking of peripherally activated lymphocytes may play a role in generating a robust intracranial immune response. Therefore, a blood-based assay to identify peripheral blood response may both predict response and better identify the ideal patient populations for future ICI clinical trials.

Objectives:

Determine if the outcomes, as measured by overall survival, is improved in patients with newly diagnosed glioblastoma when treatment with immune checkpoint inhibitors result in an immune response in peripheral blood T lymphocytes.

Eligibility:

Histologically confirmed, newly diagnosed primary glioblastoma or gliosarcoma;

Age greater than or equal to 18 years;

Adequate organ function;

Karnofsky performance score greater than or equal to 70;

Subjects must recently complete resection and chemoradiation;

Subjects must not have prior immunotherapy, other current investigational agents, or corticosteroid treatment > 30mg cortisone-equivalents per day.

Design:

Open-label, investigator-initiated exploratory study of newly-diagnosed GBM who have completed resection and chemoradiation.

Participants will be randomized to be treated in Arm 1 or 2, consistent of adjuvant chemotherapy (temozolomide (TMZ)) and immunotherapy (nivolumab + ipilimumab):

TMZ (150-200 mg/m2 PO on days 1-5 q28 days for cycles 1-6)

Arm 1:

Nivolumab (1 mg/kg IV q2weeks for cycles 1-4, then 480 mg IV q4weeks for cycles 5-16) + ipilimumab (1 mg/kg IV q4 weeks for cycles 1-4)

Arm 2:

Nivolumab (1 mg/kg IV q2weeks for cycles 1-4, then 480 mg IV q4weeks for cycles 5-16) + ipilimumab (3 mg/kg IV q4 weeks for cycles 1-4)

For the primary objective, serial examination of peripheral blood, including comprehensive flow cytometric analysis of leukocyte populations and cytokines, and Interferon- >= (IFN- >=) ELISPOT functional analysis of CD4+/8+ response to common recall antigens will be used to determine systemic response to ICI treatment.

For the secondary objectives, correlative studies assess peripheral blood T cells' ability to respond to an in vitro stimulation paradigm, including nivolumab and ipilimumab, in a microbead-based model. The T cell response to pretreatment in vitro stimulation would be compared to post-treatment in vivo stimulation to determine if this in vitro model can predict in vivo response.

Additional exploratory studies are planned to characterize the in vivo immune response to adjuvant chemotherapy and immunotherapy, including but not limited to:

Phospho-flow functional analysis of NK cell response to IFN/IL-15 stimulation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have newly diagnosed histologically confirmed primary glioblastoma or gliosarcoma
* Participants must have undergone an extensive resection of unifocal, confined to the supratentorial compartment, tumor.
* Participant must have completed chemoradiation (external beam radiation with concurrent temozolomide) a maximum of 5 weeks prior to initiation of study therapy. Potential participants who have a limited short term, reversable, unrelated to their underlying disease, concurrent illness, the initiation of treatment may be delayed up to 14 days, if the participant meet all other I/E criteria at that time.
* Age greater than or equal to 18 years.
* Karnofsky greater than or equal to 70%
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/mcL
  * Platelet Count >100,000/mcL
  * Hemoglobin > 9.0 g/dL (may be transfused to achieve this level)
  * BUN less than or equal to 30 mg/dL
  * Serum creatinine less than or equal to 1.7 mg/dL or creatinine clearance as measured by 24 hour urine collection as > 60 ml/min.
  * Total bilirubin (except participants with Gilbert s Syndrome, who are eligible for the study but exempt from the total bilirubin eligibility criterion) less than or equal to 2.0 mg/dL
  * ALT and AST less than or equal to 2.5x institutional upper limit of normal.
* The effects of study treatment on the developing human fetus are unknown. For this reason, participants of reproductive potential must agree to abstinence or use adequate contraception which includes a combination of TWO of the following:

  * Barrier method of contraception: condoms (male or female) with or without a spermicidal agent, diaphragm, or cervical cap with spermicide
  * IUD
  * Hormone-based contraceptive
  * Tubal ligation

Note: Consider use in individuals of child-bearing potential (IOCBP) only or both individuals who can father children and IOCBP starting from the enrollment and for the duration of study treatment and up to 6 months (IOCBP) after the last dose of study drug and 6 months (if individual can father children) after the last dose of temozolomide. Should a IOCBP become pregnant or suspect pregnancy while the individual or partner is participating in this study, the individual should inform the treating physician immediately.

-The participant must be able to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Definitive clinical or radiologic evidence of progressive disease.
* Prior placement of Gliadel wafer or local brachytherapy. Note: Tumor Treating Fields are allowed.
* Participants who are receiving any other investigational agents.
* Participants who have a history of receiving immune therapy, such as a vaccine therapy, dendritic cell vaccine or intracavitary or convectional enhanced delivery of therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, ipilimumab or temozolomide.
* History of allergic reactions attributed to gadolinium contrast.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Prior or concurrent malignancy unless its natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Participants with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These include but are not limited to participants with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome or CIDP, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease

(IBD), Crohn s, ulcerative colitis, and hepatitis; and participants with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome. Such diseases should be excluded because of the risk of recurrence or exacerbation of disease.

Note: Participants with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Participants with rheumatoid arthritis and other arthropathies, Sjogren s syndrome, psoriasis controlled with topical medication, and participants with positive serology, such as antinuclear antibodies (ANA) and anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.

* The participant must not be currently on a corticosteroid dose greater than physiologic replacement dosing defined as 30 mg of cortisone per day or its equivalent. Participants must have stopped corticosteroids above this threshold at least 7 days prior to initiation of study treatment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations (within timeframes identified in the bullets below) that

would limit compliance with study requirements.

* Individual who are pregnant are excluded from this study because study treatment potential for teratogenic or abortifacient effects is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to study treatment of the mother, breastfeeding should be discontinued.
* Known active, chronic, or history of hepatitis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine if the outcomes, as measured by overall survival, is improved in patients with newly diagnosed glioblastoma when treatment with immune checkpoint inhibitors result in an immune response in peripheral blood T lymphocytes. | death
  Correlation between the Median amount of time subject survives after therapy and quantitative analysis of peripheral blood T lymphocytes.

SECONDARY OUTCOMES:
Determine if the T cell response measured by the ex vivo tosylactivated bead assay correlates with subsequent systemic response to treatment with immune checkpoint inhibitors. | Baseline, Day 1 of each Cycle and 60 day and 100 day post treatment
  Correlation between T cell response to immune checkpoint inhibitors and survival
Determine if T cell response to immune checkpoint inhibitors measuring the change in the pre-treatment and post-treatment blood correlates with progression-free survival | disease progression
  Measurement of pretreatment and posttreatment blood correlates and its correlation T cell response to checkpoint inhibitors.
Determine if in vitro peripheral blood T cell response to a stimulation paradigm including nivolumab and ipilimumab correlates with progression-free survival, evaluating 2 different dosing regimens of the ICIs. | disease progression
  Correlation between T cell response with varying dose regimen of immune checkpoint inhibitors and disease progression
Determine if in vitro peripheral blood T cell response to a stimulation paradigm including nivolumab and ipilimumab correlates with overall survival, evaluating 2 different dosing regimens of the ICIs. | death
  Correlation between T cell response with varying dose regimen of immune checkpoint inhibitors and death
Evaluate changes in patient reported outcome measures using self-reported symptom severity and interference with daily activities using the MDASI-BT with treatment response and progression-free and overall survival. | Study Calendar, last collection of QOL Questioner
  Proportion of patients that have an improvement in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
BTRIS: All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@CTA: All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: BTRIS: Clinical data available during the study and indefinitely.@@@@@@All collected IPD will be available after primary analysis have been published.
Access Criteria: BTRIS: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2021-C-0015.html